CLINICAL TRIAL: NCT06343415
Title: Intensive Gait-assisted Versus Intensive Step-assisted Training After Acquired Brain Injury - a Randomised Cross-over Feasibility Trial.
Brief Title: Robot-assisted Training After Acquired Brain Injury and Disorders of Consciousness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christina Kruuse (Other)
Responsible Party: Sponsor-Investigator, Christina Kruuse, Professor, Dr Med, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: H-23052844
Record Dates: First submitted 2024-03-14; First posted 2024-04-02 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Acquired Brain Injury; Disorders of Consciousness
Keywords: Brain injury; Traumatic brain injury; consciousness; robot-assisted gait training; tilt-table; feasibility; cross-over study
MeSH Terms: conditions — Brain Injuries; Consciousness Disorders; Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: AB - BA
Who Masked: Outcomes Assessor
Masking Description: Assessors are blinded to allocation for the following exploratory clinical outcome scales: "Disability Rating Scale" and "Coma Recovery Scale-Revised".
  Data analyses are blinded by coding and blinding the groups (groups A and B) for the statistical analyses. After the analysis, two separate conclusions will be written before lifting the blinding and revealing the results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GAIT-assisted training (Active Comparator): Gait-assisted training in the Lokomat Pro, (Hocoma, Switzerland) for five consecutive days. The Lokomat Pro is a fully automated robotic training device consisting of a treadmill, a body weight support system, two motor-driven leg orthoses, a screen for augmented feedback and a therapist-controlled computer.
  The orthoses drive the swing phase of the gait, and their guidance force is adjusted between 10-100%. The body weight support can be adjusted between 10-100% of the body weight. The maximum walking speed is 3 km/h, and the cadence of the orthoses is calibrated to the treadmill.
  The Lokomat has five different emergency and safety stops. Every 5 minutes, an automatic signal reminds the therapist to check in; if not, the Lokomat will automatically stop. Only therapist that has gone through specific education can operate the Lokomat.
  Interventions: Other: GAIT-assisted training
- STEP-assisted training (Active Comparator): Step-assisted training in the Erigo Pro, (Hocoma, Switzerland) for five consecutive days.
  The computer-controlled tilt table consists of a verticalization table up to 90° and a choice of cyclic leg movements in three distinct patterns, between 8-80 steps/minute adjustable between 0-100% guidance force. The tilt table can be used with functional electric stimulation (FES). Weight-bearing of the legs is possible between 0-50 kg.
  The Erigo has one safety stop and an emergency release handle in case of a power failure during operation. Only therapist that has gone through specific introduction can operate the Erigo.
  Interventions: Other: STEP-assisted training

INTERVENTIONS:
Other: GAIT-assisted training — GAIT duration starts when walking is started. The participant will walk as intensively as possible within prespecified safety limits. Intensity is considered the most important factor for the feasibility outcome of the completion ratio and for the safety outcomes. Intensity encompasses duration and repetitions.
  Duration: 10 minutes is considered the minimum acceptable duration for a session to be deemed complete and 30 minutes as the maximum duration for a training session.
  Repetitions: A step intensity of approximately 1000 steps per session is considered as high intensity and training aims to reach this amount. This is based on neuroplasticity theories. Speed starts at 1 km/h and is adjusted accordingly.
  The body weight support (BWS) is kept between 60-100% of total body weight. The BWS is adjusted so the knee flexion in the stance phase does not exceed 10 degrees. The guidance force is kept at 100% and symmetric in all sessions.
  Other Names: Intensive gait-assisted training, Lokomat Pro
  Arms: GAIT-assisted training
Other: STEP-assisted training — STEP duration starts when stepping and elevation are started. The participant will step as intensively as possible within prespecified safety limits. Intensity is considered the most important factor for the feasibility outcome of the completion ratio and for the safety outcomes. Intensity encompasses duration and repetitions.
  Duration: 10 minutes is considered the minimum acceptable duration for a session to be deemed complete and 30 minutes as the maximum duration for a training session.
  Repetitions: A step intensity of approximately 1000 steps per session is considered as high intensity and training aims to reach this amount. This is based on neuroplasticity theories. Step cadence starts at 40 steps/minute and cadence is adjusted accordingly.
  The leg loading starts a 5 kg and is, if possible, increased to a maximum of 40% of total body weight while adjusting knee extension to ≤10 degrees flexion in stance. The guidance force is kept at 100% and symmetric in all sessions.
  Other Names: Intensive step-assisted training, Erigo Pro
  Arms: STEP-assisted training

SUMMARY:
The goal of this randomised cross-over feasibility trial is to investigate two intensive robot-assisted training therapies in the early rehabilitation phase after acquired brain injury and disorders of consciousness. The main questions it aims to answer are:

* Is the protocol feasible concerning inclusion in the study?
* Is the protocol feasible concerning protocol completion? Participants will randomly be assigned to either five days of robot-assisted gait training (GAIT), two days of pause, then five days of robot-assisted step training (STEP) or vice versa.

The investigators will explore and compare safety events, physiological measures and physical activity levels, behavioural measures, and functional disability outcomes. Further, the investigators report intervention and technical parameters in detail.

DETAILED DESCRIPTION:
This is a randomised cross-over feasibility trial, carried out according to the Helsinki Declaration and approved by the scientific ethics committee of the Capital Region, Denmark. Participants are temporarily unable to consent why this obtained from the next of kin.

Participants start the intervention when 10 minutes of standing in a tilt-table does not cause orthostatic hypotension. Participants then recieve five days of intervention, two days pause and then cross over to the other intervention.

Groups:

1. GAIT --> STEP
2. STEP --> GAIT

ELIGIBILITY:
INCLUSION CRITERIA

* Admitted for rehabilitation at the Department of Brain and Spinal Cord Injury, Division of Brain Injury, Bodil Eskesen Centre, Rigshospitalet
* Patients 18 years or older
* In the unresponsive wakefulness or minimally conscious state after a moderate to severe acquired brain injury (ICD 10: S06, Intracranial injury; I60-I69, Cerebrovascular diseases)
* Obtained consent from nearest relative and study guardian.

EXCLUSION CRITERIA

* Weight > 135 kg (maximum weight for the Erigo® tilt table)
* Height > 200 cm (maximum height for the Lokomat®)
* In the confusional state or emerged to full consciousness
* If weight bearing is restricted due to, e.g., fractures of the spine, pelvis, or lower limbs.
* Known osteoporosis of a severity where use of robotic orthoses, according to a physician, is considered a contraindication
* If lower limb joints are fixated to a degree that cannot be compensated in the orthoses
* No valid consent from the nearest relative or study guardian

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Inclusion Rate | 26 days from intervention start
  To be deemed feasible, the inclusion rate must be 70% (12 out of 17 eligible patients), with a 95% confidence interval (CI) from 46.9% to 86.7%.
  The data analyses are blinded by coding and blinding the groups (groups A and B) for the statistical analyses. After the analysis, two separate conclusions will be written before lifting the blinding and revealing the results.
Completion Ratio of protocols | 26 days from intervention start
  To be deemed feasible, the ratio of completed sessions must be 80% (68 out of 85 sessions per group) with a 95% CI from 70.3% to 87.1%.
  The data analyses are blinded by coding and blinding the groups (groups A and B) for the statistical analyses. After the analysis, two separate conclusions will be written before lifting the blinding and revealing the results.

SECONDARY OUTCOMES:
Exploratory Safety Outcomes | 26 days from intervention start
  Adverse events and reactions are recorded during, between and after interventions (days 1 to 26).

OTHER OUTCOMES:
Disability Rating Scale (DRS) | 26 days from intervention start
  The DRS assesses the overall disability in patients with brain injuries in 8 functional areas in 4 categories. The scores range between 0 (no disability) to 29 (extreme vegetative state). A clinician performs the test, which requires no specific training, and takes about 15 minutes or can be done by interviewing staff or relatives. The assessment is blinded for allocation.
Coma Recovery Scale-Revised (CRS-R) and level of consciousness | 26 days from intervention start
  The CRS-R assesses the level of consciousness in patients with acquired brain injury and is used for monitoring the course of recovery. It consists of 6 subscales, and the scoring is based on specific behavioural responses to standardised sensory stimuli at the bedside. The minimum score is 0 (reflexive activity), and the maximum score is 23 (cognitively mediated behaviour). A trained clinician performs the test, which takes 15-30 minutes to administer. The CRS-R has a high sensitivity for detecting signs of consciousness and includes criteria for both minimally conscious state and emergence, plus and minus. A score of 10 or greater indicates a minimally conscious state or the emergence minimally conscious state. A trained neuropsychologist blinded for allocation performs the CRS-R.
Early Functional Abilities (EFA) | 26 days from intervention start
  The EFA assesses the functional status in the early stages of recovery after acquired brain injury. It comprises 20 items in 5 subscales rated on a 5-point ordinal scale. The minimum score is 20 (no function), and the maximum score is 100 (normal function). The EFA has been shown to have a ceiling effect with better functioning. The scoring is based on observations within the last 72 hours and takes 15-30 minutes to administer. The patient's team administers the EFA why assessment is not blinded to allocation.
Functional Independence Measure (FIM) | 26 days from intervention start
  The FIM assesses the severity of disability in rehabilitation patients and how much assistance is required for an individual to perform activities of daily living. It consists of 18 items (13 motor tasks and five cognitive tasks) rated on a 7-point ordinal scale. Scores range from 18 (totally dependent) to 126 (completely independent). The FIM has some floor effects in patients with low function. The scoring is based on observations within the last 72 hours and takes 15-30 minutes to perform the scale. The patient's team administers the FIM why assessment is not blinded to allocation.
Physical activity intensity | during intervention period (10 days) during training sessions
  The investigators explore if GAIT and STEP induce a cardiovascular response resembling physical activity, even though muscular activity might be absent. The percentage of heart rate max (HRmax) is used as an indicator of physical activity intensity.
  HRmax is calculated from the following formulas:
  Female: HRmax = 209.273 - 0.803 x age (R2 = 0.55) Male: HRmax = 208.609 - 0.716 x age (R2 = 0.47)
  "Physical activity intensity" is reported using the following cut-offs for physical activity levels: Light intensity: < 65% of HRmax. Moderate intensity: 65-75% of HRmax. Vigorous intensity: 76-96% of HRmax.
  In addition, the time (minutes) spent in light, moderate, or vigorous physical activity is explored.
Mean arterial pressure (MAP) | during intervention period (10 days), after training sessions
  The mean arterial pressure is, among others, regulated by the baroreceptors. It is explored how blood pressure regulates after GAIT and STEP. Continuous non-invasive arterial pressure (CNAP) and MAP are measured in a resting position before GAIT/STEP preparation. The investigators measure CNAP and MAP after the training session when the patient is positioned in a resting position (sitting or lying.)
Heart Rate Variability (HRV) | during intervention period (10 days), end of intervention
  The HRV is suggested to reflect responsiveness in patients with disorders of consciousness indirectly. HRV might reflect the interaction between the autonomic nervous system and cognitive, sensory, behavioural, and affective processes. The HRV is also an indirect measure of the sympathetic/parasympathetic balance. The HRV signal is obtained from the heart rate measures; the high frequency (HF) interval reflects parasympathetic activity (0.15-0.5Hz; HF); the low-frequency (LF) interval reflects mainly sympathetic but also parasympathetic activity (0.04-0.015 Hz; LF) and is typically correlated to physical stress; The LF/HF is classically considered an index of "sympathetic- vagal balance" of heart rate regulation, particularly during long-term recordings and is thus classically an expression of the baroreceptor feedback loop. It is expected that the interventions stimulate patient awakeness and awareness, which might be reflected in a change in HRV.
Behavioural Outcome | First and last session of each arm (30 minutes, 4 sessions per participant)
  It is investigated if behavior differ between interventions. Behavior can be either random/not goal oriented, or a response/goal oriented to an input. This is evaluated from video recordings from the first and last session of each intervention where behavior like communication, visual awareness, and motor output are analysed.
  Behavioural changes are explored from observations not blinded to allocation.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Kruuse, Professor, Study Director — Rigshospitalet, Denmark
Locations (1):
- Department of brain and spinal cord injury, Glostrup Municipality, Greater Copenhagen, Denmark